CLINICAL TRIAL: NCT04415047
Title: A Study to Assess Safety and Effectiveness of the JenaValve Trilogy™ Heart Valve System in the Treatment of High Surgical Risk Patients With Symptomatic, Severe Aortic Regurgitation (AR)
Brief Title: The JenaValve ALIGN-AR Pivotal Trial
Acronym: ALIGN-AR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02C320
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Aortic Regurgitation; Aortic Valve Insufficiency; Aortic Insufficiency; Aortic Valve Disease
Keywords: Valvular Heart Disease; Aortic Incompetence; Aortic Valve Incompetence
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Disease; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcatheter Aortic Valve Replacement (TAVR) (Experimental): TAVR with JenaValve Trilogy Heart Valve System Intervention Device: JenaValve Trilogy Heart Valve System
  Interventions: Device: JenaValve Trilogy Heart Valve System

INTERVENTIONS:
Device: JenaValve Trilogy Heart Valve System — TAVR with JenaValve Trilogy Heart Valve System

SUMMARY:
To collect information about treatment for symptomatic severe Aortic Regurgitation (AR), which affects the aortic valve in the heart. Aortic regurgitation is a condition where aortic valve in the heart does not close tightly and allows some blood to leak back into the heart chamber. Symptoms of aortic regurgitation may include fatigue and shortness of breath. The preferred treatment for severe aortic regurgitation is aortic valve replacement surgery.

DETAILED DESCRIPTION:
This study will examine the use of TAVR (Transcatheter Aortic Valve Replacement), which is a minimally invasive procedure designed to replace the aortic valve inside the heart. In this study, TAVR will be performed using the JenaValve Pericardial TAVR System, which is intended to help treat symptomatic severe aortic regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe aortic regurgitation (AR).
* Patient at high risk for open surgical valve replacement
* Patient symptomatic according to NYHA functional class II or higher
* The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB)/ Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

* Congenital uni or bicuspid aortic valve morphology
* Previous prosthetic aortic valve (bioprosthesis or mechanical) implant
* Endocarditis or other active infection
* Need for urgent or emergent TAVR procedure for any reason
* Cardiogenic shock or hemodynamic instability requiring inotropic support or ventricular assist device
* Severe mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-08-29 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality at 1 Year | 1 year
  All-cause mortality within the first 12 months post index procedure
All Stroke | 30 days
  Number of patients that had a stroke
Major Bleeding | 30 days
  Number of patients that had any of these events
Acute Kidney Injury | 30 days
  Number of patients that had these events
Major Vascular Complications | 30 days
  Number of patients that had these events
Surgery/intervention related to the device | 30 days
  Number of patients that had these events
Permanent pacemaker implantation | 30 days
  Number of patients that had these events
Total aortic regurgitation | 30 days
  Number of patients that had these events

SECONDARY OUTCOMES:
KCCQ | 1 year
  KCCQ Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, MD, Study Chair — New York-Presbyterian/ Columbia University Medical Center; Torsten P. Vahl, MD, Principal Investigator — New York-Presbyterian/ Columbia University Medical Center; Vinod H. Thourani, MD, Principal Investigator — Piedmont Healthcare
Locations (30):
- United States (30):
  - TMC HealthCare & PIMA Heart, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Scripps Hospital, San Diego, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant/ BayCare Health, Clearwater, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Cardiac Surgery Clinical Research Center Inc./ Advocate Aurora Health, Oak Lawn, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute/ Abbott Northwestern, Minneapolis, Minnesota
  - Barnes-Jewish Hospital / Washington University, St Louis, Missouri
  - Rutgers Robert Wood Johnson Medical School/ Rutgers Robert Wood University Hospital, Piscataway, New Jersey
  - New York-Presbyterian/ Columbia University Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Allegheny-Singer Health Network, Pittsburgh, Pennsylvania
  - Lankenau, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Memorial Hermann - Texas Medical Center, Houston, Texas
  - Intermountain Medical Center Heart Institute, Salt Lake City, Utah
  - Sentara Hospitals, Norfolk, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoghbi WA, Adams D, Bonow RO, Enriquez-Sarano M, Foster E, Grayburn PA, Hahn RT, Han Y, Hung J, Lang RM, Little SH, Shah DJ, Shernan S, Thavendiranathan P, Thomas JD, Weissman NJ. Recommendations for Noninvasive Evaluation of Native Valvular Regurgitation: A Report from the American Society of Echocardiography Developed in Collaboration with the Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr. 2017 Apr;30(4):303-371. doi: 10.1016/j.echo.2017.01.007. Epub 2017 Mar 14. No abstract available. PMID 28314623
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Jun 20;135(25):e1159-e1195. doi: 10.1161/CIR.0000000000000503. Epub 2017 Mar 15. No abstract available. PMID 28298458
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Geyer M, Tamm AR, Munzel T, Treede H, von Bardeleben RS. Novel Transfemoral TAVR System to Treat Aortic Regurgitation in Degenerated Surgical Aortic Valve Replacement Even in Unfavorable Anatomy. JACC Cardiovasc Interv. 2022 Jun 13;15(11):e135-e136. doi: 10.1016/j.jcin.2022.02.043. Epub 2022 May 11. No abstract available. PMID 35568645
- [Background] Poschner T, Werner P, Kocher A, Laufer G, Musumeci F, Andreas M, Russo M. The JenaValve pericardial transcatheter aortic valve replacement system to treat aortic valve disease. Future Cardiol. 2022 Feb;18(2):101-113. doi: 10.2217/fca-2021-0065. Epub 2021 Oct 14. PMID 34647465
- [Background] Ng VG, Khalique OK, Nazif T, Patel A, Hamid N, George I, Bapat V, Hahn R, Kodali S, Vahl TP. Treatment of Acute Aortic Insufficiency With a Dedicated Device. JACC Case Rep. 2021 Mar 24;3(4):645-649. doi: 10.1016/j.jaccas.2021.01.021. eCollection 2021 Apr. PMID 34317595
- [Derived] Makkar RR, Thourani VH, Vahl TP, Yadav PK, McCabe JM, George I, Satler L, Chetcuti S, Daniels DV, Waggoner T, Whisenant B, Russo M, Summers M, Garcia S, Frisoli T, Ramana RK, Stinis C, Golwala H, Zahr F, Greenbaum A, Rovin J, Sanchez C, Szerlip M, Deeb GM, Amoroso N, Patel D, Fahy M, Ranard LS, Gupta A, Chakravarty T, Skaf S, Chuang M, Kodali SK, Figulla HR, Treede H, Baldus S, Pinto DS, Leon MB; ALIGN-AR Investigators. Transcatheter aortic valve implantation with the Trilogy valve for symptomatic native aortic regurgitation (ALIGN-AR): a pivotal, multicentre, single-arm, investigational device exemption study. Lancet. 2025 Dec 13;406(10521):2757-2771. doi: 10.1016/S0140-6736(25)02215-9. Epub 2025 Nov 16. PMID 41260228
- [Derived] Vahl TP, Thourani VH, Makkar RR, Hamid N, Khalique OK, Daniels D, McCabe JM, Satler L, Russo M, Cheng W, George I, Aldea G, Sheridan B, Kereiakes D, Golwala H, Zahr F, Chetcuti S, Yadav P, Kodali SK, Treede H, Baldus S, Amoroso N, Ranard LS, Pinto DS, Leon MB. Transcatheter aortic valve implantation in patients with high-risk symptomatic native aortic regurgitation (ALIGN-AR): a prospective, multicentre, single-arm study. Lancet. 2024 Apr 13;403(10435):1451-1459. doi: 10.1016/S0140-6736(23)02806-4. Epub 2024 Mar 26. PMID 38552656
- [Derived] Hamid N, Ranard LS, Khalique OK, Hahn RT, Nazif TM, George I, Ng V, Leon MB, Kodali SK, Vahl TP. Commissural Alignment After Transfemoral Transcatheter Aortic Valve Replacement With the JenaValve Trilogy System. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2079-2081. doi: 10.1016/j.jcin.2021.07.025. No abstract available. PMID 34556282